CLINICAL TRIAL: NCT05861544
Title: Pomegranate Juice Consumption by Patients Under Medication for Addiction Treatment as a Regulator of Craving and Blood Redox Status: The Study Protocol of a Randomized Control Trial (the NUTRIDOPE Study)
Brief Title: NUTRItion-driven Detoxification of OPioid Addicted patiEnts
Acronym: NUTRIDOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Organization Against Drugs (ΟΚΑΝΑ) (Other Government)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Christonikos Leventelis, Toxicologist, MSc, PhD, Organization Against Drugs (ΟΚΑΝΑ)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 44482-2/12/2020
Record Dates: First submitted 2023-04-13; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Psychiatry
Keywords: Craving; Buprenorphine; Opioid use disorders; Methadone; Pomegranate juice; Redox biomarkers; Inflammation; Antioxidants; Nutrition
MeSH Terms: conditions — Opioid-Related Disorders; Inflammation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients under medication for addiction treatment (MAT) that are active members of the Greek Organization Against Drugs (OKANA) therapeutic units will be recruited for this investigation. The participants will be stratified into two subgroups, i.e., methadone maintenance treatment (MMT) and buprenorphine maintenance treatment (BMT), according to the maintenance treatment program they attend. Pomegranate juice, which is the examined nutritional intervention, will be administered to the participants of both MMT and BMT subgroups of the experimental group. The juice will be administered to the patients at the following dosage: 250 ml/day, seven days/week, for four months.
  Interventions: Dietary Supplement: Pomegranate juice
- Control group (No Intervention): Patients under medication for addiction treatment (MAT) that are active members of the Greek Organization Against Drugs (OKANA) therapeutic units under methadone or buprenorphine treatment. The participants will be stratified into two subgroups, i.e., methadone maintenance treatment (MMT) and buprenorphine maintenance treatment (BMT), according to the maintenance treatment program they attend. The patients of the control group (both MMT and BMT subgroups) will not consume any similar beverage as a placebo due to the objective difficulties of making one that will be identical to the fresh pomegranate juice.

INTERVENTIONS:
Dietary Supplement: Pomegranate juice — The pomegranate juice that will be used in the experiment is a 100% natural product without conservatives. It will kindly be donated from the company Rodi Hellas SA, Pella, Greece. The product is in line with the quality assurance certificates by the International Organization for Standardization (ISO 22000:2005), Global Gap, Grasp and Kosher.
  Arms: Experimental group

SUMMARY:
The NUTRIDOPE (NUTRItion-driven Detoxification of OPioid addicted patiEnts) study is a clinical trial that aims to investigate the role of pomegranate juice consumption by opioid-addicted patients under buprenorphine and methadone on craving, which is the primary outcome, and other parameters. In detail, fresh pomegranate juice will be administered for 120 days (250 ml, 7 days/week) to the patients and craving as well as other psychosocial (e.g., depression, mood state, quality of life) and biochemical (i.e., blood redox status and inflammation) parameters will be evaluated. It is hypothesized that pomegranate juice will reduce craving probably through the improvement of blood redox and inflammation status.

Pomegranate juice, which is the examined nutritional intervention, will be administered to the participants of the experimental group, whereas their counterparts in the control group will not consume any similar beverage as a placebo due to the objective difficulties of making one that will be identical and not separable with the fresh pomegranate juice.

DETAILED DESCRIPTION:
Background: Buprenorphine and methadone are considered the "gold standard" medication for addiction treatment (MAT) for patients with opioid use disorders (OUDs). However, they may cause side effects promoting craving (i.e., opioid use relapse). Therefore, the concurrent administration of natural products could be an adjunct intervention to back up opioid MAT. Pomegranate is a natural substance that contains antioxidant polyphenolic compounds, which have been associated with craving reduction. Moreover, pomegranate positively affects psychosocial parameters, such as depression and anxiety that are common feelings for patients with OUDs, probably due to its potent antioxidant and anti-inflammatory properties.

Objectives: The NUTRIDOPE (NUTRItion-driven Detoxification of OPioid addicted patiEnts) study aims to investigate the role of pomegranate juice consumption by patients with OUDs under buprenorphine and methadone on craving.

Methods: Fresh pomegranate juice will be administered for 120 days (250 ml, 7 days/week) and craving, as the primary outcome, as well as other psychosocial (e.g., depression, mood state, quality of life) and biochemical (i.e., blood redox status and inflammation) parameters will be evaluated.

Anticipated Results: It is hypothesized that pomegranate juice will reduce craving probably through the improvement of blood redox and inflammation status.

Conclusions: NUTRIDOPE is a hypothesis-driven, evidence-based, multifactorial project that proposes a nutrition-based solution towards craving reduction for patients with OUDs under MAT, potentially assisting towards their successful rehab and societal reintegration.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years of age
* Long-term heroin or other opioid drug use
* Suffering from physical and mental dependence due to chronic opioid use

Exclusion Criteria:

* Serious medical problems, such as infection by human immunodeficiency virus or hepatitis B virus
* Current use of anti-inflammatory medication
* Relapse to other addictive substances (i.e., opioids, methamphetamine, benzodiazepines, cannabis, tetrahydrocannabinol, amphetamine) - To rule out the use of such substances, all participants underwent weekly urine tests during the four-month period of the experiment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-07-23 (Estimated); Study Completion 2024-01-23 (Estimated)

PRIMARY OUTCOMES:
Craving | Changes between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement) will be assessed.
  Heroin Craving Questionnaire (HCQ), which is a validated instrument, will be used for the assessment of the effects of pomegranate juice on craving. It is consisted of 45 questions divided in 5 dimensions, namely desire to use heroin, intentions and planning to use heroin, anticipation of positive outcome, relief from withdrawal or dysphoria, and lack of control overuse. HCQ will be completed by the volunteers of both the experimental and control groups at four timepoints in order to assess the change on craving as follows: Before the start of the experiment (i.e., day 1 or baseline), in the middle of the experiment (i.e., day 60), at the end of the experiment (i.e., day 120), and 6 months after the end of the experiment (i.e., follow-up measurement).

SECONDARY OUTCOMES:
Quality of Life (QoL) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  The Nottingham Health Profile (NHP) questionnaire will be used for the assessment of the pomegranate juice effects on the QoL of the patients. The questionnaire consists of two parts; the first part assesses parameters such as activity, pain, emotional reaction, sleep, social isolation, and mobility, whereas the second part evaluates the effects of health or disease on the activities of daily living.
Determination of antioxidant enzyme Catalase (CAT) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Spectrophotometric evaluation of the activity of the antioxidant enzyme CAT expressed in U/gr Hb (haemoglobin) in red blood cell lysate (RBCL). The enzyme activity will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the total antioxidant capacity (TAC) of plasma | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  TAC will be evaluated spectrophotometrically in plasma expressed as mmol DPPH•/ml. TAC levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
In vitro evaluation of antioxidant and reducing properties of the administered pomegranate juice | Day 1
  The antioxidant and reducing properties of pomegranate juice will be evaluated using specific in vitro tests: 2,2-diphenyl-1-picrylhydrazyl (DPPH), 2,2'-azino-bis(3-ethylbenzothiazoline-6-sulfonic acid) (ABTS), hydroxyl radical, superoxide radical, Fe+3 to Fe2+ reduction) expressed in half maximal inhibitory concentration (IC50) (μl).
Measurement of the concentration of protein carbonyls | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Protein carbonyls, as a biomarker of protein oxidation, will be evaluated in plasma spectrophotometrically expressed in nmol/mg protein. The levels of protein carbonyls will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the concentration of thiobarbituric acid reactive substances (TBARS) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  TBARS, a biomarker of lipid peroxidation, will be evaluated in plasma spectrophotometrically expressed in μmol/l. The levels of TBARS will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the capacity of plasma to reduce hydroxyl radical (OH•) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Spectrophotometric evaluation of the ability of plasma to reduce hydroxyl radical expressed in mmol deoxyribose/ml. The reducing capacity of plasma will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the capacity of plasma to reduce superoxide radical (O2•-) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Spectrophotometric evaluation of the ability of plasma to reduce superoxide radical expressed in % scavenging capacity. The reducing capacity of plasma will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the reducing power | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Spectrophotometric evaluation of the ability of plasma to reduce Fe+3 to Fe+2 expressed in mmol potassium ferricyanide/ml. The reducing capacity of plasma will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of GSH concentration | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  The reduced form of glutathione (GSH) as a crucial antioxidant molecule will be measured spectrophotometrically and its levels will be expressed in μmol/g Hb. GSH levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the activity of the antioxidant enzyme superoxide dismutase (SOD) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  The activity of the antioxidant enzyme SOD expressed in U/gr Hb (haemoglobin) will be measured in red blood cell lysate (RBCL). SOD activity levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the activity of the antioxidant enzyme glutathione peroxidase (GPx) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  The activity of the antioxidant enzyme GPx expressed in U/gr Hb (haemoglobin) will be measured in red blood cell lysate (RBCL). GPx activity levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the activity of the antioxidant enzyme glutathione reductase (GR) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  The activity of the antioxidant enzyme GR expressed in U/gr Hb (haemoglobin) will be measured in red blood cell lysate (RBCL). GR activity levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the concentration of interferon gamma (IFN-γ) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  IFN-γ, expressed in pg/ml, is a cytokine that recruits macrophages at the site of inflammation. Its concentration will be assessed through immunofluorescence. IFN-γ levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the concentration of interferon alpha-2 (IFN-a2) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  IFN-a2, expressed in pg/ml, regulates the activation of the immune system and inhibits cell proliferation. Its concentration will be assessed through immunofluorescence. IFN-a2 levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the concentration of interleukin-1 betta (IL-1b) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  IL-1b, expressed in pg/ml, is activated by macrophages and neutrophils and regulate immune response. Its concentration will be assessed through immunofluorescence. IL-1b levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the concentration of interleukin-8 (IL-8) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Chemokine IL-8, expressed in pg/ml, induces chemotaxis of neutrophils and other granulocytes in an inflammation site. Its concentration will be assessed through immunofluorescence. IL-8 levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the concentration of monocyte chemoattractant protein-1 (MCP-1) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  MCP-1,expressed in pg/ml, recruits monocytes, lymphocytes, and neutrophils at the site of inflammation. Its concentration will be assessed through immunofluorescence. MCP-1 levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the concentration of interleukin-1 alpha (IL-1a) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  IL-1a, expressed in pg/m, regulates immune response after its activation by macrophages and neutrophils. Its concentration will be assessed through immunofluorescence. IL-1a levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the concentration of tumor necrosis factor alpha (TNF-a) | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  TNF-a, expressed in pg/ml, is realised by macrophages for cell signaling as part of the immune response. Its concentration will be assessed through immunofluorescence. TNF-a levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the concentration of melatonin | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Melatonin is involved in circadian regulation through sleep-wake timing. Saliva samples will be taken at 22.00 in dim light by patients themselves under oral and typed guidelines. Dim light melatonin onset (DLMO) concentration will be measured using enzyme-linked immunosorbent assay (ELISA) and will be expressed in pg/ml. Melatonin levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Measurement of the concentration of cortisol | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Cortisol belongs to glycocorticoid class of hormones related with stress system and can weaken the activity of immune system through the releasing of cytokines in inflammation site. Plasma samples will be collected early in the morning and cortisol concentration will be expressed in pg/ml and be measured using enzyme-linked immunosorbent assay (ELISA). Cortisol levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).

OTHER OUTCOMES:
Sleep evaluation | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Pittsburgh Sleep Quality Index (PSQI) self-reported questionnaire assesses through a Likert scale from 0-3 sleep quality and quantity, sleep habits related to quality and occurrence of sleep disturbances in adults consisting of seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. A score is calculated by the sum of the 7 components ranging between 0 and 21. The quality of sleep will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Fatigue evaluation | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Fatigue Severity Scale (FSS) is a 9-item, self-administered questionnaire which assesses the magnitude of fatigue that the patients have experienced throughout the past weeks. Fatigue levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Mood | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Profile of Mood States (POMS-short version) questionnaire consists of 37 self-administered items and assesses current mood states in 6 dimensions, namely tension, depression, anger, vigour, fatigue, and confusion. Mood levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Evaluation of constipation | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Patient Assessment of Constipation - Quality of Life (PAC-QOL) questionnaire consists of 28 self-reported items that assess the effects of constipation on the patient QOL during the last two weeks. It comprises four dimensions referring to physical discomfort, psychosocial discomfort, treatment satisfaction and worries discomfort. The responses are scored on a Likert scale ranging from 0 to 5. Higher score indicates increase of severity of the negative effects of the intervention in question on QOL. Constipation levels will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).
Faecal evaluation | Day 1; Day 60; Day 120, six months following the end of the experiment (follow-up measurement)
  Bristol Stool Form Scale (BSFS) will be used as a pictorial representation of each stool type ranging from the hardest (i.e., type 1) to the softest (i.e., type 7) related to specific bowel symptoms, such as constipation. Faecal evaluation will be compared between Day 1 (baseline) and the following time points: Day 60, Day 120, six months following the end of the experiment (follow-up measurement).

CONTACTS AND LOCATIONS:
Overall Officials: Christonikos Leventelis, Dr, Principal Investigator — Organization against Drugs
Locations (1):
- Organization Against Drugs, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this investigation will be provided to qualified researchers with related academic interest.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting one year after article publication and the data will be made accessible for up to 24 months.
Access Criteria: Access to trial data can be requested by qualified researchers and will be provided following review and approval research approval.

REFERENCES:
- [Background] Abu-Taweel GM, Al-Mutary MG. Pomegranate juice moderates anxiety- and depression-like behaviors in AlCl3-treated male mice. J Trace Elem Med Biol. 2021 Dec;68:126842. doi: 10.1016/j.jtemb.2021.126842. Epub 2021 Aug 17. PMID 34418746
- [Background] Adams LS, Seeram NP, Aggarwal BB, Takada Y, Sand D, Heber D. Pomegranate juice, total pomegranate ellagitannins, and punicalagin suppress inflammatory cell signaling in colon cancer cells. J Agric Food Chem. 2006 Feb 8;54(3):980-5. doi: 10.1021/jf052005r. PMID 16448212
- [Background] Adel-Mehraban MS, Tansaz M, Mohammadi M, Yavari M. Effects of pomegranate supplement on menopausal symptoms and quality of life in menopausal women: A double-blind randomized placebo-controlled trial. Complement Ther Clin Pract. 2022 Feb;46:101544. doi: 10.1016/j.ctcp.2022.101544. Epub 2022 Feb 2. PMID 35134697
- [Background] Ahmadi J, Jahromi MS, Ghahremani D, London ED. Single high-dose buprenorphine for opioid craving during withdrawal. Trials. 2018 Dec 10;19(1):675. doi: 10.1186/s13063-018-3055-z. PMID 30526648
- [Background] Aliyu IM, Danladi S, Ibrahim UI, Al-kassim Hassan M, Rohin MAK and Mohamad N (2018) Therapeutic potential of pomegranate antioxidant compounds in ameliorating opiate addiction. The Pharma Innovation Journal 7(5): 668-672.
- [Background] Brown R, Kraus C, Fleming M, Reddy S. Methadone: applied pharmacology and use as adjunctive treatment in chronic pain. Postgrad Med J. 2004 Nov;80(949):654-9. doi: 10.1136/pgmj.2004.022988. PMID 15537850
- [Background] Browne CJ, Godino A, Salery M, Nestler EJ. Epigenetic Mechanisms of Opioid Addiction. Biol Psychiatry. 2020 Jan 1;87(1):22-33. doi: 10.1016/j.biopsych.2019.06.027. Epub 2019 Jul 8. PMID 31477236
- [Background] Cambay Z, Baydas G, Tuzcu M, Bal R. Pomegranate (Punica granatum L.) flower improves learning and memory performances impaired by diabetes mellitus in rats. Acta Physiol Hung. 2011 Dec;98(4):409-20. doi: 10.1556/APhysiol.98.2011.4.4. PMID 22173022
- [Background] Chen SL, Lee SY, Tao PL, Chang YH, Chen SH, Chu CH, Chen PS, Lee IH, Yeh TL, Yang YK, Hong JS, Lu RB. Dextromethorphan attenuated inflammation and combined opioid use in humans undergoing methadone maintenance treatment. J Neuroimmune Pharmacol. 2012 Dec;7(4):1025-33. doi: 10.1007/s11481-012-9400-1. Epub 2012 Sep 19. PMID 22990619
- [Background] Dunn KE, Finan PH, Andrew Tompkins D, Strain EC. Frequency and correlates of sleep disturbance in methadone and buprenorphine-maintained patients. Addict Behav. 2018 Jan;76:8-14. doi: 10.1016/j.addbeh.2017.07.016. Epub 2017 Jul 14. PMID 28735039
- [Background] Estrada-Camarena EM, Lopez-Rubalcava C, Ramirez-Rodriguez GB, Pulido D, Cervantes-Anaya N, Azpilcueta-Morales G, Granados-Juarez A, Vega-Rivera NM, Islas-Preciado D, Trevino S, de Gortari P, Gonzalez-Trujano ME, Garcia-Viguera C. Aqueous extract of pomegranate enriched in ellagitannins prevents anxiety-like behavior and metabolic changes induced by cafeteria diet in an animal model of menopause. Neurochem Int. 2020 Dec;141:104876. doi: 10.1016/j.neuint.2020.104876. Epub 2020 Oct 10. PMID 33049337
- [Background] Fahmy HA, Farag MA. Ongoing and potential novel trends of pomegranate fruit peel; a comprehensive review of its health benefits and future perspectives as nutraceutical. J Food Biochem. 2022 Jan;46(1):e14024. doi: 10.1111/jfbc.14024. Epub 2021 Dec 19. PMID 34923641
- [Background] Garratt M, Brooks RC. A genetic reduction in antioxidant function causes elevated aggression in mice. J Exp Biol. 2015 Jan 15;218(Pt 2):223-7. doi: 10.1242/jeb.112011. Epub 2014 Dec 18. PMID 25524980
- [Background] Guerrero-Solano JA, Jaramillo-Morales OA, Velazquez-Gonzalez C, De la O-Arciniega M, Castaneda-Ovando A, Betanzos-Cabrera G, Bautista M. Pomegranate as a Potential Alternative of Pain Management: A Review. Plants (Basel). 2020 Mar 30;9(4):419. doi: 10.3390/plants9040419. PMID 32235455
- [Background] Hajipour S, Sarkaki A, Mohammad S, Mansouri T, Pilevarian A, RafieiRad M. Motor and cognitive deficits due to permanent cerebral hypoperfusion/ischemia improve by pomegranate seed extract in rats. Pak J Biol Sci. 2014 Aug;17(8):991-8. doi: 10.3923/pjbs.2014.991.998. PMID 26031017
- [Background] Leventelis C, Goutzourelas N, Kortsinidou A, Spanidis Y, Toulia G, Kampitsi A, Tsitsimpikou C, Stagos D, Veskoukis AS, Kouretas D. Buprenorphine and Methadone as Opioid Maintenance Treatments for Heroin-Addicted Patients Induce Oxidative Stress in Blood. Oxid Med Cell Longev. 2019 Apr 9;2019:9417048. doi: 10.1155/2019/9417048. eCollection 2019. PMID 31093318
- [Background] Lu RB, Wang TY, Lee SY, Chen SL, Chang YH, See Chen P, Lin SH, Chu CH, Huang SY, Tzeng NS, Lee IH, Chin Chen K, Kuang Yang Y, Chen P, Chen SH, Hong JS. Correlation between interleukin-6 levels and methadone maintenance therapy outcomes. Drug Alcohol Depend. 2019 Nov 1;204:107516. doi: 10.1016/j.drugalcdep.2019.06.018. Epub 2019 Aug 30. PMID 31513981
- [Background] Luvian-Morales J, Varela-Castillo FO, Flores-Cisneros L, Cetina-Perez L, Castro-Eguiluz D. Functional foods modulating inflammation and metabolism in chronic diseases: a systematic review. Crit Rev Food Sci Nutr. 2022;62(16):4371-4392. doi: 10.1080/10408398.2021.1875189. Epub 2021 Jan 28. PMID 33506690
- [Background] Mansouri MT, Naghizadeh B, Ghorbanzadeh B. Ellagic acid enhances morphine analgesia and attenuates the development of morphine tolerance and dependence in mice. Eur J Pharmacol. 2014 Oct 15;741:272-80. doi: 10.1016/j.ejphar.2014.08.024. Epub 2014 Aug 30. PMID 25179576
- [Background] Mohd Adnan LH, Mohamad N, Che Mat K, Abu Bakar NH, Hashim SN and Mohd Shariff MH (2018) Attenuation of morphine-induced cAMP overshoot by thymoquinone in opioid receptor expressing cells (U87 MG) mediated by chronic morphine treatment. Journal of Engineering and Applied Sciences.13: 8906-8911.
- [Background] Morvaridzadeh M, Sepidarkish M, Daneshzad E, Akbari A, Mobini GR, Heshmati J. The effect of pomegranate on oxidative stress parameters: A systematic review and meta-analysis. Complement Ther Med. 2020 Jan;48:102252. doi: 10.1016/j.ctim.2019.102252. Epub 2019 Nov 22. PMID 31987244
- [Background] Paur R, Wallner C, Hermann P, Stollberger C, Finsterer J. Neurological abnormalities in opiate addicts with and without substitution therapy. Am J Drug Alcohol Abuse. 2012 May;38(3):239-45. doi: 10.3109/00952990.2011.644001. Epub 2012 Jan 20. PMID 22263960
- [Background] Perrotti LI, Weaver RR, Robison B, Renthal W, Maze I, Yazdani S, Elmore RG, Knapp DJ, Selley DE, Martin BR, Sim-Selley L, Bachtell RK, Self DW, Nestler EJ. Distinct patterns of DeltaFosB induction in brain by drugs of abuse. Synapse. 2008 May;62(5):358-69. doi: 10.1002/syn.20500. PMID 18293355
- [Background] Pujol CN, Paasche C, Laprevote V, Trojak B, Vidailhet P, Bacon E, Lalanne L. Cognitive effects of labeled addictolytic medications. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Feb 2;81:306-332. doi: 10.1016/j.pnpbp.2017.09.008. Epub 2017 Sep 14. PMID 28919445
- [Background] Ridzwan N, Jumli MN, Baig AA, Rohin MAK. Pomegranate-derived anthocyanin regulates MORs-cAMP/CREB-BDNF pathways in opioid-dependent models and improves cognitive impairments. J Ayurveda Integr Med. 2020 Oct-Dec;11(4):478-488. doi: 10.1016/j.jaim.2019.12.001. Epub 2020 May 16. PMID 32430240
- [Background] Salarian A, Kadkhodaee M, Zahmatkesh M, Seifi B, Bakhshi E, Akhondzadeh S, Adeli S, Askari H, Arbabi M. Opioid Use Disorder Induces Oxidative Stress and Inflammation: The Attenuating Effect of Methadone Maintenance Treatment. Iran J Psychiatry. 2018 Jan;13(1):46-54. PMID 29892317
- [Background] Sangi S, Ahmed SP, Channa MA, Ashfaq M, Mastoi SM. A new and novel treatment of opioid dependence: Nigella sativa 500 mg. J Ayub Med Coll Abbottabad. 2008 Apr-Jun;20(2):118-24. PMID 19385474
- [Background] Sani IH, Sulaiman I, Zubairu I, Abdussalam US and Adzim MKR (2018) Antioxidant Potential of Phoenix dactylifera Linn Extract and its Effects on Calcium Channel Antagonist in the Treatment of Withdrawal Syndrome in Morphine Dependent Rats. Tropical Journal of Natural Product Research. 2(7): 309-313.
- [Background] Sason A, Adelson M, Schreiber S, Peles E. The prevalence of constipation and its relation to sweet taste preference among patients receiving methadone maintenance treatment. Drug Alcohol Depend. 2021 Aug 1;225:108836. doi: 10.1016/j.drugalcdep.2021.108836. Epub 2021 Jun 24. PMID 34182372
- [Background] Veskoukis AS, Kerasioti E, Priftis A, Kouka P, Spanidis Y, Makri S and Kouretas D (2019) A battery of translational biomarkers for the assessment of the in vitro and in vivo antioxidant action of plant polyphenolic compounds: the biomarker issue. Current Opinion in Toxicology 13: 99-109.
- [Background] Wang P, Zhang Q, Hou H, Liu Z, Wang L, Rasekhmagham R, Kord-Varkaneh H, Santos HO, Yao G. The effects of pomegranate supplementation on biomarkers of inflammation and endothelial dysfunction: A meta-analysis and systematic review. Complement Ther Med. 2020 Mar;49:102358. doi: 10.1016/j.ctim.2020.102358. Epub 2020 Feb 26. PMID 32147056
- [Derived] Leventelis C, Makri S, Ververi A, Papageorgiou K, Tentolouri A, Mountzouridi E, Tekos F, Barmpas PT, Tasoulis S, Metsios GS, Kouretas D, Veskoukis AS. Pomegranate juice ameliorates craving and oxidative stress on patients under medication for opioid addiction treatment with methadone and buprenorphine: A ranzomised controlled trial. Clin Nutr ESPEN. 2025 Apr;66:34-45. doi: 10.1016/j.clnesp.2025.01.025. Epub 2025 Jan 10. PMID 39798867